CLINICAL TRIAL: NCT00828256
Title: Outcome Study of Arthroscopic Repair of Chronic Rotator Cuff Tears Between 2005-2008, at the Soroka University Medical Center, Beer Sheva, Israel
Brief Title: Outcome of Arthroscopic Repair of Chronic Rotator Cuff Tears Between 2005-2008
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Dr. Asaf Acker, Soroka University Medical Center, Beer Sheva, Israel
Other Study IDs: sor477308ctil; isrctn9930305
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Rotator Cuff Tear
Keywords: arthroscopic repair; rotator cuff; tears; shoulder; chronic tear of rotator cuff
MeSH Terms: conditions — Rotator Cuff Injuries; Lacerations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

INTERVENTIONS:
Procedure: arthroscopy of shoulder — arthroscopic repair of chronic rotator cuff tears

SUMMARY:
Arthroscopic repair has become the preferable surgical technique to treat rotator cuff tears in the last decade. Many researches demonstrate equal and even superior outcome with this surgical technique, while others show opposite results.

The aim of this study is to estimate the anatomic and functional results of the arthroscopic repair among the patients of the orthopedic department at the Soroka University Medical Center, in order to check the investigators hypothesis that indeed - the arthroscopic repair of the rotator cuff is the better surgical technique.

Methods: study population - 80 patients who had had an arthroscopic repair of the rotator cuff between the years 2005-2008 at the SUMC.

Inclusion criteria: age over 18 years. arthroscopic rotator cuff repair. date of operation not before 2005.

Study design:

1. Data base Collection.
2. Inviting the patients for physical examination + ultrasound examination of the operated shoulder + filling out questionnaires (SF36, CONSTANT SCORE)
3. Statistical analysis
4. Publication

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Arthroscopic repair of chronic rotator cuff tear
* Operation done after January 2005

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 patients, above 18 years of age, who had had an arthroscopic repair of chronic rotator cuff tear between the years 2005-2008.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-05 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
evidence of an anatomic repair of the rotator cuff proved by ultrasound | immidiate

SECONDARY OUTCOMES:
high constant score | 6 months after surgery